CLINICAL TRIAL: NCT07330453
Title: Early Prediction and Clinical Outcomes of Cardiovascular Surgery-Associated Acute Kidney Injury: A Prospective Multicenter Cohort Study
Brief Title: Cardiovascular Surgery Early Prediction System for AKI :CARDS-AKI Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Sheng Liu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2025ZD0547500
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Surgery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Perioperative Blood and Urine Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who did not develop acute kidney injury(AKI) after cardiovascular surgery
  Interventions: Other: Observation
- Patients who developed AKI after cardiovascular surgery
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — As an observational study, patients' therapeutic approach will not be modified during the course of this research.

SUMMARY:
This multicenter, prospective study prospectively enrolled patients undergoing cardiovascular surgery. Detailed perioperative clinical data and biospecimens were collected at multiple time points. The primary aim is to develop an early warning model for postoperative acute kidney injury (AKI) by integrating clinical data and biomarkers. Additionally, through long-term follow-up, the study seeks to characterize outcome trajectories and establish a prognostic model for AKI patients.

This study addresses four key questions: 1) Integration of clinical information and biomarkers to develop an early predictive model for cardiac surgery-associated acute kidney injury (CSA-AKI); 2) Identification of risk factors for CSA-AKI occurrence; 3) Determinants of prognosis in patients with CSA-AKI; and 4) Enhanced prediction of near- and long-term clinical event risks in this patient population.

Participants will receive standard perioperative management. The study protocol includes the following procedures:(1) Clinical Data Collection: Comprehensive perioperative clinical data will be systematically recorded. (2) Biospecimen Sampling: Serial blood and urine samples will be obtained at predefined time points throughout the perioperative period. (3) In-Hospital Monitoring: Clinical outcomes will be continuously monitored during the hospital stay. (3) Post-discharge Follow-up: Participants will be assessed at regular intervals after discharge to track the occurrence of major adverse events.

These findings provide a foundational basis for the development of a data-driven early-warning system. Such a system is designed to facilitate the prompt identification of high-risk patients and enable the initiation of personalized treatment strategies, thereby potentially improving clinical outcomes and optimizing resource allocation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years；
* Scheduled to undergo elective cardiac surgery；
* Able to complete baseline data collection and provide written informed consent.

Exclusion Criteria:

* Preoperative serum creatinine > 353 μmol/L, history of or currently receiving dialysis therapy.
* History of kidney transplantation.
* Presence of malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fuwai Hospital, CAMS & PUMC, Peking University People's Hospital; Guangdong People's Hospital; Fuwai Hospital Shenzhen (Sun Yat-sen Cardiovascular Hospital, Shenzhen); Huaxi Hospital, Sichuan University; Yantai Yuhuangding Hospital; Fuwai Centarl China Cardiovascular Hospital; Fuwai Yunnan Hospital, Academy of Medical Science; Yinzhou District Center for Disease Control and Prevention, Ningbo; Peking University First Hospital
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of post-operative acute kidney injury | From the end of surgery to 48 hours postoperative

SECONDARY OUTCOMES:
The occurrence of adverse kidney events up to 2 years. | 2 years
The occurrence of adverse cardiovascular events up to 2 years. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided